CLINICAL TRIAL: NCT03199820
Title: Prostaglandin Insert (Propess) Versus Trans-cervical Balloon Catheter for Out-patient Labour Induction: A Randomised Controlled Trial of Feasibility
Brief Title: Balloon Catheter Versus Propess for Labour Induction
Acronym: PROBIT-F
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St George's, University of London (Other)
Collaborators: City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13.0029
Record Dates: First submitted 2017-05-31; First posted 2017-06-27 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Childbirth Problems; Labor Complication
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial of feasibility
Who Masked: Outcomes Assessor
Masking Description: The trial statistician will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cook Cervical balloon (Active Comparator): Cook cervical double balloon catheter
  Interventions: Device: Cook cervical balloon
- Prostin E2 Vaginal suppository (Active Comparator): Prostaglandin E2 sustained release vaginal insert
  Interventions: Drug: Prostin E2 Vaginal Suppository

INTERVENTIONS:
Device: Cook cervical balloon — trans-cervical balloon catheter for out-patient labour induction
  Arms: Cook Cervical balloon
Drug: Prostin E2 Vaginal Suppository — Propess Vaginal suppository for out-patient Labour induction
  Other Names: Propess
  Arms: Prostin E2 Vaginal suppository

SUMMARY:
This study will randomise low-risk women to compare the effectiveness of trans-cervical balloon catheter for pre-induction cervical ripening for out-patient induction of labour with current practice (Propess). Women will be randomised to two treatment groups. The investigators wish to explore if such a trial is feasible, acceptable to women and what data collection is required for a future trial. Since no data exist, the investigators propose a study with approximately 60 women in each arm across two recruiting sites.

DETAILED DESCRIPTION:
The study will be conducted over two sites: St. George's Hospital in London, and Medway Hospital in Kent. Women requiring induction of labour (IOL) at term will be invited to participate in the study, where they will be randomised to either the trans-cervical balloon catheter or the vaginal prostaglandin 10mg (Propess).

Consent to enter this study will be obtained after 37+0 weeks after a full account has been provided of its nature, purpose, risks, burdens and potential benefits. Patients will have the opportunity to consider whether they wish to take part in the study, up to a maximum of 72 hours. For prolonged pregnancy (41+0 weeks), Induction of labour is generally booked at 41+3 weeks, giving a 3-day time period to think about participation. Periods shorter than 72 hours will be permitted if the woman felt that further deliberation will not lead to a change in her decision, and provided the person seeking consent is satisfied that the woman has fully retained, understood and deliberated on the information given. This provision has been made with the support of our patient advisory group. Likewise, periods longer than 72 hours will be permitted should the woman request this. The Investigator or designee will explain that the women are under no obligation to enter the trial and that they can withdraw at any time during the trial, without having to give a reason. A copy of the signed Informed Consent Form will be given to the study participant. The original signed consent form (ICF) will be retained at the study site in the Investigation site file (ISF) and a copy of the ICF along with a copy of the Participant Information Sheet (PIS) will be retained in the maternity notes.

If new safety information results in significant changes to the risk-benefit assessment, the consent form will be reviewed and updated if necessary. All subjects, including those already treated, will be informed of the new information, given a copy of the revised consent form and asked to re-consent if they choose to continue in the study.

In order to ensure a similar distribution between treatment groups in important characteristics thought to affect outcomes, including site and parity, allocation will be random and stratified by site (St. George's and Medway) and parity (nulliparous and multiparous). Participants will be allocated using block randomisation so as to ensure similar numbers of participants in the treatment groups. Whilst blocks of size four are proposed, advice regarding random block sizes (including four, six and eight) will be sought from the Kings Clinical Trials Unit (CTU).

Participants and midwives will not be blinded to the treatment allocation. The trial statistician will be blinded to group allocation.

The trial will be analysed using an intention to treat approach. Induction of labour with Propess: 10mg insert will be introduced in the posterior vaginal fornix close to the cervix as recommended by the manufacturer. Women will undergo monitoring of fetal condition and uterine activity by cardio-tocography (CTG) according to the existing protocol. It will be discontinued once the CTG is deemed to be normal. The woman will be allowed home with instructions to return to the hospital at an agreed time, 18-24 hours later, or if in labour, whichever was earlier. On the following morning the pessary will be removed, and artificial rupture of membranes (ARM) attempted.

Induction of labour with balloon catheter: The woman should be positioned in the lithotomy position and insert a large vaginal speculum to gain cervical access. The cervix must be cleaned appropriately to prepare for device insertion. Insert the device into the cervix and advance until both balloons have entered the cervical canal. Inflate the uterine balloon with 40ml Sodium Chloride (NaCL) 0.9% using a standard luer lock 20ml syringe through the red check-flo valve marked U.

Once the uterine balloon is inflated, the device is pulled back until the balloon is against the internal cervical os. The vaginal balloon is now visible outside the external cervical os. Inflate the vaginal balloon with 20ml NaCl 0.9% using a standard luer lock 20ml syringe through the green Check-Flo valve marked V. Once the balloons are situated on each side of the cervix and the device is fixed in place, remove the speculum. Add more fluid to each balloon in turn, in 20ml increments until each balloon contains 80ml (maximum volume of fluid) Do NOT overinflate the balloons. If desired the end of the catheter may be taped to the woman's thigh.

Women will undergo monitoring of fetal condition and uterine activity by cardio-tocography (CTG) according to the existing protocol. It will be discontinued when the CTG is deemed to be normal. The woman will be allowed home with instructions to return to the hospital an agreed time, 18-24 hours later, or if in labour, whichever was earlier. When the participant returns, the balloon catheter will be removed, and artificial rupture of membranes (ARM) attempted.

If artificial rupture of membranes was not possible, this will be considered as treatment failure and alternative ways of achieving delivery will be sought as per local guidelines and followed. Unsuccessful placement of the balloon or inability to perform ARM will be considered as treatment failure and an alternative method of IOL will be used.

Survey

1. Recruitment Survey. Questionnaires will be given to all women at the point of recruitment. Women who decline will be invited to complete the questionnaire anonymously and it will be made clear that the aim of the survey is solely to improve future care through assessing the feasibility of the balloon catheter with no implications for their own care. The schedule will comprise closed questions plus comment boxes to examine women's understanding of the trial, their reasons for participation or declining. A detailed process log will also be maintained to identify the numbers and proportions of women who accept randomisation and those who withdraw after entry to the trial.
2. Follow-up questionnaire for participants: We will use a slightly modified form of questionnaire used previously used by Henry et al (2013) to assess patient satisfaction, experience of participating, experience of the IoL process using either method including pain or discomfort, experience of outpatient IoL and level of information provided.

Qualitative study In addition, qualitative data will be gathered for a sample of participants to enable a fuller exploration of the trial feasibility in two stages.

1. To gain a better understanding of feasibility and effective trial procedures for a trial where interventions cannot be blinded and preferences may be strong. A researcher with experience of studies of trial processes, independent of the trial management, will (with consent of women and professionals) observe a sample of recruitment discussions to ascertain how information is provided and to understand in greater depth how choices about trial participation are made. The focus will include diversity issues, as typically participation in randomized controlled trials (RCTs) is socially and ethnically skewed. This will be a consecutive sample continued until saturation to include women allocated randomly and those in the preference arms, those women who decline and a cross-section of social and ethnic groups. Estimated sample: 40 recruitment observations.
2. Women included in observations who consented to participate in the trial will be invited to participate in semi structured interviews postnatally, to explore their experience of participating and of the IoL process using either method, their experience of outpatient IOL and any further reflections. Those who provide telephone details will be contacted postnatally to confirm whether they are still happy to participate in an interview, following checks of neonatal outcomes. All women and professionals will be assured of confidentiality and their rights to decline consent for observation or interview. A thematic framework analysis will be conducted focused on lessons for trial feasibility, design, recruitment and retention, and patient experiences of cervical ripening using either method for induction in an outpatient setting. This approach enables consideration of unintended as well as anticipated consequences plus a fuller understanding of how women and their birth partners experience induction of labour and whether an outpatient approach confers advantages in terms of experience and satisfaction since, despite this being a key rationale for an outpatient approach, patient experiences of different induction approaches is an under-explored area. The number of interviews will be guided by data saturation, with a maximum potential sample of 40.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women with a single fetus and uncomplicated pregnancy, with a gestational age > 37+ 0 weeks, needing induction of labour

1. ≥18 years of age
2. No medical risk factors.

Exclusion Criteria:

1. Out-patient induction of labour is deemed unsuitable for the following women on the grounds of safety -

   * Grand multiparous women (Parity 5 or more)
   * Multiple pregnancy
   * Women with complex medical or obstetric problems (i.e. placenta previa, recurrent antepartum hemorrhage, diabetes, pre-eclampsia, Intrauterine growth restriction (UGR), Obstetric Cholestasis)
   * Previous caesarean section/uterine scar
2. Women who are contracting and/ or requiring analgesia
3. Women who do not fully understand the information leaflet and unable to provide full informed consent
4. Women for whom out-patient induction is unsuitable according to local hospital protocol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 120 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
feasibility of randomised Induction of Labour Trial in Out-patient setting | 12 months
  Number of eligible women willing to enrol

CONTACTS AND LOCATIONS:
Overall Officials: Amarnath Bhide, MD, Principal Investigator — St. George's University Hospitals Foundation Trust
Locations (2):
- United Kingdom (2):
  - Medway Maritime Hospital, Gillingham, Kent
  - St Georges University Hospital NHS Foundation Trust, Tooting, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kelly AJ, Alfirevic Z, Ghosh A. Outpatient versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2013 Nov 12;(11):CD007372. doi: 10.1002/14651858.CD007372.pub3. PMID 24222365
- [Result] Dowswell T, Kelly AJ, Livio S, Norman JE, Alfirevic Z. Different methods for the induction of labour in outpatient settings. Cochrane Database Syst Rev. 2010 Aug 4;(8):CD007701. doi: 10.1002/14651858.CD007701.pub2. PMID 20687092
- [Result] Henry A, Madan A, Reid R, Tracy SK, Austin K, Welsh A, Challis D. Outpatient Foley catheter versus inpatient prostaglandin E2 gel for induction of labour: a randomised trial. BMC Pregnancy Childbirth. 2013 Jan 29;13:25. doi: 10.1186/1471-2393-13-25. PMID 23356673
- [Result] Pennell CE, Henderson JJ, O'Neill MJ, McChlery S, Doherty DA, Dickinson JE. Induction of labour in nulliparous women with an unfavourable cervix: a randomised controlled trial comparing double and single balloon catheters and PGE2 gel. BJOG. 2009 Oct;116(11):1443-52. doi: 10.1111/j.1471-0528.2009.02279.x. Epub 2009 Jul 28. PMID 19656148
- [Result] Jozwiak M, Oude Rengerink K, Benthem M, van Beek E, Dijksterhuis MG, de Graaf IM, van Huizen ME, Oudijk MA, Papatsonis DN, Perquin DA, Porath M, van der Post JA, Rijnders RJ, Scheepers HC, Spaanderman ME, van Pampus MG, de Leeuw JW, Mol BW, Bloemenkamp KW; PROBAAT Study Group. Foley catheter versus vaginal prostaglandin E2 gel for induction of labour at term (PROBAAT trial): an open-label, randomised controlled trial. Lancet. 2011 Dec 17;378(9809):2095-103. doi: 10.1016/S0140-6736(11)61484-0. Epub 2011 Oct 24. PMID 22030144
- [Result] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Result] Wilkinson C, Bryce R, Adelson P, Turnbull D. A randomised controlled trial of outpatient compared with inpatient cervical ripening with prostaglandin E(2) (OPRA study). BJOG. 2015 Jan;122(1):94-104. doi: 10.1111/1471-0528.12846. Epub 2014 May 14. PMID 24824157
- [Result] Howard K, Gerard K, Adelson P, Bryce R, Wilkinson C, Turnbull D. Women's preferences for inpatient and outpatient priming for labour induction: a discrete choice experiment. BMC Health Serv Res. 2014 Jul 30;14:330. doi: 10.1186/1472-6963-14-330. PMID 25073486
- [Result] Hannah ME, Hannah WJ, Hewson SA, Hodnett ED, Saigal S, Willan AR. Planned caesarean section versus planned vaginal birth for breech presentation at term: a randomised multicentre trial. Term Breech Trial Collaborative Group. Lancet. 2000 Oct 21;356(9239):1375-83. doi: 10.1016/s0140-6736(00)02840-3. PMID 11052579
- [Result] Turnbull D, Adelson P, Oster C, Coffey J, Coomblas J, Bryce R, Wilkinson C. The impact of outpatient priming for induction of labour on midwives' work demand, work autonomy and satisfaction. Women Birth. 2013 Sep;26(3):207-12. doi: 10.1016/j.wombi.2013.03.001. Epub 2013 Apr 3. PMID 23561927
- [Result] O'Brien E, Rauf Z, Alfirevic Z, Lavender T. Women's experiences of outpatient induction of labour with remote continuous monitoring. Midwifery. 2013 Apr;29(4):325-31. doi: 10.1016/j.midw.2012.01.014. Epub 2012 Nov 16. PMID 23159160
- [Result] Norman JE, Stock S. Intracervical Foley catheter for induction of labour. Lancet. 2011 Dec 17;378(9809):2054-5. doi: 10.1016/S0140-6736(11)61581-X. Epub 2011 Oct 24. No abstract available. PMID 22030142
- [Result] Ten Eikelder ML, Oude Rengerink K, Jozwiak M, de Leeuw JW, de Graaf IM, van Pampus MG, Holswilder M, Oudijk MA, van Baaren GJ, Pernet PJ, Bax C, van Unnik GA, Martens G, Porath M, van Vliet H, Rijnders RJ, Feitsma AH, Roumen FJ, van Loon AJ, Versendaal H, Weinans MJ, Woiski M, van Beek E, Hermsen B, Mol BW, Bloemenkamp KW. Induction of labour at term with oral misoprostol versus a Foley catheter (PROBAAT-II): a multicentre randomised controlled non-inferiority trial. Lancet. 2016 Apr 16;387(10028):1619-28. doi: 10.1016/S0140-6736(16)00084-2. Epub 2016 Feb 3. PMID 26850983
- [Result] Wilkinson C, Adelson P, Turnbull D. A comparison of inpatient with outpatient balloon catheter cervical ripening: a pilot randomized controlled trial. BMC Pregnancy Childbirth. 2015 May 28;15:126. doi: 10.1186/s12884-015-0550-z. PMID 26018581
- [Derived] Scamell M, Meades R, Foya V. Embodiment and the technologies of induction of labour. Midwifery. 2024 Nov;138:104144. doi: 10.1016/j.midw.2024.104144. Epub 2024 Aug 14. PMID 39232460
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Bhide A, Sedgwick P, Barrett B, Cupples G, Coates R, Goode R, Linton S, McCourt C. Prostaglandin insert dinoprostone versus trans-cervical balloon catheter for outpatient labour induction: a randomised controlled trial of feasibility (PROBIT-F). Pilot Feasibility Stud. 2020 Aug 15;6:113. doi: 10.1186/s40814-020-00661-7. eCollection 2020. PMID 32821419